CLINICAL TRIAL: NCT02944500
Title: Saxenda: Underlying Mechanisms and Clinical Outcomes
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2015P000327
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Brain; Liraglutide; MRI
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide followed by placebo (Experimental): Participants will receive liraglutide with dose titration over 5 weeks (0.6mg for 1 week, 1.2mg for 1 week, 1.8mg for 1 week, 2.4mg for 1 week, and 3.0mg for 1 week) followed by a minimum of 3 weeks wash-out and then return for the same dose of placebo for the same amount of time.
  Interventions: Drug: liraglutide; Other: Placebo
- Placebo followed by liraglutide (Experimental): Participants will receive placebo with dose titration (0.6mg for 1 week, 1.2mg for 1 week, 1.8mg for 1 week, 2.4mg for 1 week, and 3.0mg for 1 week) followed by a minimum of 3 weeks wash-out and then return for the same dose of liraglutide for the same amount of time.
  Interventions: Drug: liraglutide; Other: Placebo

INTERVENTIONS:
Drug: liraglutide
  Other Names: Saxenda
Other: Placebo

SUMMARY:
The purpose of this protocol is to investigate the effect of treatment with the study drug Liraglutide, a GLP-1 receptor agonist, on centers of the brain that control appetite and food intake.

DETAILED DESCRIPTION:
The effect of treatment with the study drug Liraglutide, a recently discovered GLP-1 receptor agonist, on centers of the brain that control appetite and food intake will be studied in detail.

ELIGIBILITY:
Inclusion Criteria:

* Obese: BMI> 30 kg/m2 or >27 kg/m2 with comorbidities (including but not limited to insulin resistance, hypertension, dyslipidemia, cardiovascular disease, stroke, sleep apnea, gallbladder disease, hyperuricemia and gout, and osteoarthritis).

Exclusion Criteria:

1. Women who are breastfeeding, pregnant, or wanting to become pregnant.
2. Women using metal IUD
3. Any change in the dosage of hormonal contraceptive medications (birth control pills, implanon). Subjects should remain on same medication/ same dose during the time of the entire study.
4. Moderate (creatinine clearance of 30-59 ml/min) and severe renal impairment (creatinine clearance below 30 ml/min) and end-stage renal disease
5. Moderate, or severe hepatic impairment
6. Hypersensitivity to the active substance or any of the excipients in liraglutide
7. History of diabetic ketoacidosis
8. Congestive heart failure
9. EKG abnormalities (as listed above)
10. Inflammatory conditions like inflammatory bowel disease, Rheumatoid arthritis etc
11. Gastroparesis
12. Pancreatitis
13. Gallstones- as they may cause increased risk of pancreatitis
14. Alcohol consumption- the maximum quantity for men is 140g-210g per week. For women, the range is 84g-140g per week or drinking as consuming no more than two drinks a day for men and one for women. Alcohol can cause increased risk of pancreatitis and hypoglycemia.
15. Untreated thyroid disease like hypothyroidism or hyperthyroidism
16. Subjects taking the following medications: warfarin, steroids (inhaled or systemic due to reduced hypoglycemic effect), and subjects on other hormones (LHRH analogs etc).
17. Subjects on any oral anti-diabetic agent except metformin
18. Personal or family history of MEN II or medullary thyroid cancer
19. Subjects with any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neuron or biostimulators, electronic infusion pumps, etc.)
20. Subjects with any type of metallic implant that could potentially be displaced or damaged during MRI, such as aneurysm clips, metallic skull plates, surgical implants etc. or metal containing tattoos
21. Anxiety of small spaces and/or claustrophobia
22. Uncontrolled cardiac impairment, circulatory impairment, or inability to perspire (poor thermoregulatory function)
23. Significant sensory or motor impairment
24. Epilepsy, particularly photo-sensitive epilepsy, which may place the individual at a higher risk for adverse events during fMRI scanning with visual stimulation
25. Subjects with neurological or psychological problems which may interfere with or complicate testing (e.g. presence of titubation)
26. Body weight above the limitation of the MRI scanning table (330lbs/150 Kg) or body dimensions that could difficult the performance of the scan.
27. Subjects who cannot adhere to the experimental protocol for any reason
28. Anemia with Hgb less than 10
29. Uncontrolled infectious diseases (e.g. HIV, hepatitis, chronic infections etc)
30. Any uncontrolled endocrine condition, e.g Cushing's, Acromegaly, etc
31. Any cancers or lymphoma
32. Eating disorders like anorexia, bulimia
33. Severe hypertriglyceridemia (triglycerides >500 mg/dl)
34. Weight loss surgery or gastrectomy
35. Any changes in medications that affect brain function, e.g. anti-depressants, anti-psychotics, anti-anxiety, anti-seizure medications, antihypertensives etc (subjects should remain on same medication/ same dose during the time of the entire study).
36. Vegetarians- as food images presented will include numerous non-vegetarian items and thus will not be appealing as high calorie food items.
37. Suicidality, as measured by the MSSI at screening visit.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
BOLD response to food cues | 5 weeks
  effect size of BOLD response to food cues in the brain

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center General Clinical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Patient data is protected by HIPAA. Results will be published in a peer-reviewed journal.

REFERENCES:
- [Derived] Angelidi AM, Kokkinos A, Sanoudou D, Connelly MA, Alexandrou A, Mingrone G, Mantzoros CS. Early metabolomic, lipid and lipoprotein changes in response to medical and surgical therapeutic approaches to obesity. Metabolism. 2023 Jan;138:155346. doi: 10.1016/j.metabol.2022.155346. Epub 2022 Nov 12. PMID 36375643
- [Derived] Peradze N, Farr OM, Perakakis N, Lazaro I, Sala-Vila A, Mantzoros CS. Short-term treatment with high dose liraglutide improves lipid and lipoprotein profile and changes hormonal mediators of lipid metabolism in obese patients with no overt type 2 diabetes mellitus: a randomized, placebo-controlled, cross-over, double-blind clinical trial. Cardiovasc Diabetol. 2019 Oct 31;18(1):141. doi: 10.1186/s12933-019-0945-7. PMID 31672146